CLINICAL TRIAL: NCT06488430
Title: Mild Cognitive Impairment Among Community Dwelling Adults: Prevalence, Associated Factors, and Feasibility of a Multidomain Intervention Package for Preventing Cognitive Decline
Brief Title: Mild Cognitive Impairment and Multidomain Intervention Package
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); Believers Church Medical College Hospital, Tiruvalla, Kerala, India (Unknown)
Responsible Party: Principal Investigator, Vishwajit Nimgaonkar, MD PhD, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY23010015; 5D43TW009114-10 (NIH)
Record Dates: First submitted 2024-06-18; First posted 2024-07-05 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Dementia
Keywords: Dementia; cognitive ability; Mild cognitive impairment (MCI); Multidomain intervention
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Mixed-Methods study Phase 1: Quantitative design to assess the burden of mild cognitive impairment (MCI) Phase 2: Development of multidomain intervention (DONE) Phase 3: Qualitative design to explore the barriers and facilitators for adherence to intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multidomain intervention package for preventing cognitive decline (Experimental): A multidomain intervention including nutritional advice, physical activity, cognitive stimulation training, social support and engagement and management of vascular risk factors.
  Interventions: Behavioral: Multidomain intervention package for preventing cognitive decline

INTERVENTIONS:
Behavioral: Multidomain intervention package for preventing cognitive decline — Participants with mild cognitive impairment will be identified and they will participate in a pilot study for one-month duration. During pilot study they will be subjected to a multidomain intervention including nutritional advice, physical activity, cognitive stimulation training, social support and engagement and management of vascular risk factors.

SUMMARY:
The state of Kerala, India has the highest proportion of older adults and the burden of lifestyle diseases causes great concern. Therefore, there is need for identifying a feasible multidomain preventive intervention to ease this burden. Initially the burden of mild cognitive impairment will be determined as this information is scarce from the setting. A multidomain intervention package will be developed that is appropriate for the setting. The adherence rates, barriers and facilitators will be assessed. If the multidomain intervention is found feasible, it can be recommended for further clinical trials.

DETAILED DESCRIPTION:
In the context of increasing older adults, the burden of dementia is forecasted to increase in India. Interventions targeting risk factors and diseases may be the key element to counter the dementia epidemic. The state of Kerala having highest proportion of older adults and burden of lifestyle diseases in India causes even greater concern. Hence, there is need for identifying the burden of mild cognitive impairment, developing a feasible multidomain preventive intervention to be applied among older adults to prevent cognitive decline.

Objectives

1. To estimate the burden of mild cognitive impairment among community dwelling adults between 50-65 years in a taluk of a South Kerala district
2. To develop a multidomain intervention package for preventing cognitive decline in those with mild cognitive impairment

2. To explore the barriers and facilitators for adherence towards multidomain intervention to prevent cognitive decline in community dwelling older adults between 50- 65 years with mild cognitive impairment in the study area Recruitment: The sampling area consists of 54 wards (39 rural and 15 urban) from Tiruvalla Taluk of Pathanamthitta district. A ward is a division of the community at the local government level with approximately 300-500 families and an elected government representative from the community known as ward member. From these wards, 15 rural and 5 (total 20 wards) urban wards will be randomly picked. From each ward, 24 eligible participants will be randomly picked from all the wards, one extra person from the last ward in order to reach the sample size. ASHA workers will help the team to identify the eligible candidates. The ASHA workers and the ward members will communicate to the community regarding the study which would help the research team to build a rapport with the community. The research team will explain the details of the study and consent form to the potential participants. Identified, consented adults (50- to 65-year-old) will be screened using the study tool to identify those with mild cognitive impairment.

Screening: All individuals (50-65yrs) consenting to participate will be included. Those who are unable to respond, critically ill and with a diagnosis of dementia (physician diagnosed) will be excluded. MCI in the study will be assessed using the European Alzheimer's Disease Consortium. Participants who meet all the five criteria of this definition will be defined as MCI cases.

Enrollment: Twenty participants found to have MCI will be enrolled in to a pilot study to explore the barriers and facilitators of adherence towards the intervention package. The inclusion and exclusion criteria has been detailed earlier. All those with MCI from a ward will be included. If adequate number is not available in a ward, rest of the participants will be taken from the adjacent ward.

Intervention: A multidomain intervention will be developed and will be pilot tested for adherence for a period of one month. The intervention includes nutritional advice, physical activity, cognitive stimulation therapy, social engagements and, management of vascular risk factors.

Assessment The cognitive ability, depression, activities of daily living, quality of life will be assessed during the screening phase by using standard questionnaires validated in the local language. The adherence towards the individual and group activities in the intervention will be assessed using checklists. In-depth interviews will be conducted to understand the barriers and facilitators towards adherance.

Followup The research team will assess the adherence towards intervention using checklists. In depth interviews will be done to identify the barriers and facilitators towards adherence.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1- All individuals (50-65yrs) consenting to participate will be included. Phase 3- Inclusion for multidomain intervention
* Individuals between 50-65 years old, willing to participate and comply with all the study evaluation and intervention procedures
* CAIDE (Cardiovascular Risk Factors, Aging and Dementia) Dementia Risk Score of 6 points or higher
* Those identified to have mild cognitive impairment in phase 1 screening

Exclusion Criteria:

• Phase 1- Those who are unable to respond, critically ill and having a physician diagnosed dementia report will be excluded.

Phase 3- Exclusion for multidomain intervention

* Geriatric Depression Scale ≥ 9
* Dementia
* Disorders that may affect safe involvement in the intervention (eg, malignancy, symptomatic cardiovascular disease, Large vessel stroke in the past two years, History of transient ischemia attack (TIA) or small vessel stroke in the last 6 months, revascularization within 1 year previously, severe loss of vision, hearing, or communicative ability)
* Coincident participation in another intervention trial.
* Recent (< 3 months) bone fracture.
* History of hip fracture, joint replacement, or spinal surgery in the last 6 months
* Clinically significant abnormalities in laboratory blood tests as per judgment of the site study clinician.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Attention domain of Addenbrooke's Cognitive Examination-III (ACE-III). | Baseline, After one month intervention
  Change in attention domain scores of Malayalam version of Addenbrooke's Cognitive Examination (m-ACE) will be tested after intervention (Score below the cut-off in at least one of the cognitive domains assessed.
  [One SD below the mean score (of that educational category) was taken as the cut-off for each domain] The minimum score is 0 and maximum score is 18.
  )
Memory domain of Addenbrooke's Cognitive Examination-III (ACE-III). | Baseline, After one month intervention
  Change in memory domain scores of Malayalam version of Addenbrooke's Cognitive Examination (m-ACE) will be tested after intervention (Score below the cut-off in at least one of the domains tested. The lowest score is 0 and highest score is [One SD below the mean score (of that educational category) was taken as the cut-off for each domain] The minimum score is 0 and maximum score is 26.
  )
Fluency domain of Addenbrooke's Cognitive Examination-III (ACE-III). | Baseline, After one month intervention
  Change in fluency domain scores of Malayalam version of Addenbrooke's Cognitive Examination (m-ACE) will be tested after intervention (Score below the cut-off in at least one of the domains tested. The lowest score is 0 and highest score is 14.
  [One SD below the mean score (of that educational category) was taken as the cut-off for each domain] The minimum score is 0 and maximum score is 18.
  )
Language domain of Addenbrooke's Cognitive Examination-III (ACE-III). | Baseline, After one month intervention
  Change in language domain scores of Malayalam version of Addenbrooke's Cognitive Examination (m-ACE) will be tested after intervention (Score below the cut-off in at least one of the domains tested. The lowest score is 0 and highest score is 26.
  [One SD below the mean score (of that educational category) was taken as the cut-off for each domain] The minimum score is 0 and maximum score is 18.
  )
Visuospatial domain of Addenbrooke's Cognitive Examination-III (ACE-III). | Baseline, After one month intervention
  Change in visuospatial domain scores of Malayalam version of Addenbrooke's Cognitive Examination (m-ACE) will be tested after intervention (Score below the cut-off in at least one of the domains tested. The lowest score is 0 and highest score is 16.
  [One SD below the mean score (of that educational category) was taken as the cut-off for each domain] The minimum score is 0 and maximum score is 18.
  )

SECONDARY OUTCOMES:
Depression score on Geriatric Depression Scale | Baseline and after one month intervention
  Persons with dementia will be enrolled and their depression score measured. Multidomain intervention package is provided for one months and depression score is measured again. The minimum score is 0 and maximum score is 30.

CONTACTS AND LOCATIONS:
Overall Officials: Vishwajit L Nimgaonkar, MD,, Principal Investigator — university
Locations (1):
- Believers Church Medical College, Tiruvalla, Kerala, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: One year after publication of this study.
Access Criteria: For individual participant data, meta-analysis.